CLINICAL TRIAL: NCT07159061
Title: Reducing Neural Perseveration Through Closed Loop Real Time fMRI Neurofeedback to Alleviate Depressive Symptoms
Brief Title: Neurofeedback to Treat Depression - 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Yvette Sheline, McLure Professor of Radiology, Neurology and Psychiatry, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 849298-2
Record Dates: First submitted 2025-09-03; First posted 2025-09-08 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: Active Neurofeedback (Active Comparator): R33 Phase: Three training sessions. Each training session contains 32 minutes of active neurofeedback runs.
  Interventions: Behavioral: Active Closed Loop Real Time fMRI Neurofeedback
- Sham Comparator: Sham Neurofeedback (Sham Comparator): R33 Phase: Three training sessions. Each training session contains 32 minutes of sham (placebo) neurofeedback runs.
  Interventions: Behavioral: Sham Closed Loop Real Time fMRI Neurofeedback

INTERVENTIONS:
Behavioral: Active Closed Loop Real Time fMRI Neurofeedback — Active neurofeedback to target neural mechanisms underlying attentional bias in participants with major depressive discover (MDD)
  Arms: Active Comparator: Active Neurofeedback
Behavioral: Sham Closed Loop Real Time fMRI Neurofeedback — Sham (placebo) neurofeedback to target neural mechanisms underlying attentional bias in participants with major depressive discover (MDD)
  Arms: Sham Comparator: Sham Neurofeedback

SUMMARY:
This study tests the efficacy of a new psychotherapeutic strategy for reducing negative attention bias (and therefore depression severity) in participants with MDD. This real-time fMRI neurofeedback therapy uses cloud-based pattern classification to decode a patient's attentional state and dynamically modulate task stimuli (in a closed loop) based on this state.

DETAILED DESCRIPTION:
The investigators will compare cloud based real time fMRI feedback with placebo (sham feedback) in reducing negative attention bias and depressive symptoms. This study will be the first dose-finding test of real-time fMRI effect on negative attention bias. Measures include: Structured Clinical Interview for DSM-5 (SCID), Clinician-administered diagnostic exam, Montgomery Asberg Depression Rating Scale (MADRS), Clinician-administered scale used to assess the severity of depression, State-Trait Anxiety Inventory (STAI), Self-report questionnaire used to measure types of anxiety and mood symptoms, Mood and Anxiety Symptom Questionnaire (MASQ), Negative perseveration during a go/no-go task, Go/no-go task with overlaid face/scene stimuli; brain response triggers next stimulus, Negative gaze, Negative gaze collected in gaze data following each real time fMRI feedback session

ELIGIBILITY:
Inclusion Criteria:

* Gender, inclusive
* Adult aged 18 - 65
* Meets Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for MDD according to the Clinician-Administered MDD Scale for DSM-5 (unipolar depression or bipolar II depressed)
* Scores at least a minimum score of 16 on Montgomery Asberg Depression Rating Scale (MADRS)
* Normal cognition
* Participants must be able to read and understand English
* Participants must be able to provide consent

Exclusion Criteria:

* Pregnancy (female participants)
* Outside age range
* MRI contraindications (medical implant, claustrophobia, etc.)
* Use of psychoactive medication (including antidepressants) or currently in therapy
* Neurological disorder or any condition that in the view of the PI could impact brain data, cause depression, require medication that could cause depressive symptoms, or otherwise result in participant being unfit for study (for example, co-morbid psychotic, neurological disorders, developmentally or cognitively disabled/impaired, active alcohol or drug abuse/dependence within the past 6 months).
* Non-English speaking
* Non-correctable vision loss
* Refusal to provide informed consent
* representing an active suicide risk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2028-11-21 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS) | 3 months
  Clinician administered scale to assess the severity of depression. MADRS scores will be compare the effect of real-time neurofeedback vs sham neurofeedback on depression outcome in patients with MDD. A MADRS score of 16 or higher is needed in order to be eligible to be enrolled in the study. The higher the MADRS score, the more depressed the individual will be. A lower MADRS score indicates that the individual's depressive symptoms have improved. A higher MADRS score indicates that the individual's depressive symptoms have worsened.

CONTACTS AND LOCATIONS:
Overall Officials: Yvette Sheline, M.D., Principal Investigator — Center for Neuromodulation in Depression and Stress, University of Pennsylvania
Locations (1):
- Center for Neuromodulation in Depression and Stress, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Data will only be shared amongst the study sites.